CLINICAL TRIAL: NCT03881683
Title: Determination of the Feasibility of Tumoural Somatic Mutations Detection in Blood of Patients With Ovarian Cancer
Acronym: BOVARY Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-A03113-52
Record Dates: First submitted 2019-03-06; First posted 2019-03-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Ovarian Cancer
Keywords: BRCA 1/2 genes; Circulating Tumor DNA/blood*; somatic tumor mutations; HRD genes
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRD and BRCA mutations (Experimental)
  Interventions: Diagnostic Test: HRD and BRCA mutations

INTERVENTIONS:
Diagnostic Test: HRD and BRCA mutations — Compare BRCA1/2 and HRD genes mutation detected from blood sample (20 ml) and biopsy

SUMMARY:
BOVARY-Pilot is a monocentric prospective transversal pilot study with a total duration of 6 months. The purpose of this study is to determine the feasibility of detecting somatic tumor mutations in the blood of patients with ovarian cancer in order to determine whether a blood test can replace a tissue biopsy to prescribe a personalized treatment. The method will consist of a single blood sample during the patient's visit and prior to the establishment of any newly diagnosed cancer treatment. The concordance of somatic mutations (SNV) found in tissue and in cell-free DNA (cfDNA) extracted from blood will then be compared

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient with stage III to IV non-treated high grade ovarian cancer or recurrent high grade ovarian cancer
* Adequate haemoglobin rate ≥ 9 g/dL
* Patient who can benefit from an additional blood sample of 20ml. The total volume of each sample meets with the indications of the Order in force establishing the list of researches mentioned in 2 ° of Article L. 1121-1 of the Public Health Code.
* Availability of tumor samples from biopsy or surgery
* Patient affiliated to a social security scheme
* Ability to provide written informed consent

Exclusion Criteria:

* Any concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study
* Contraindication to a blood sample of 20 mL
* Pregnant or breast-feeding women
* Ongoing treatment for the newly diagnosed cancer or the recurrence
* Patient pre-treated with poly-ADP-ribose-polymérase-1 (PARP) Inhibitors
* Patient under guardianship or curatorship or deprived of liberty.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-21 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2021-02-19 (Actual)

PRIMARY OUTCOMES:
Concordance between DNA extracted from tumour tissue and cfDNA extracted from plasma (SNV, indels) | 1 day (samples will be analyzed in batch at the end of inclusions)
  Number of patients with detected punctual somatic mutations (SNVs and indels of BRCA1/2 and genes involved in HRD) concordance between DNA extracted from tumour tissue and cfDNA extracted from plasma

SECONDARY OUTCOMES:
Concordance between DNA extracted from tumour tissue and cfDNA extracted from plasma (large rearrangements, LOH, CNV) | 1 day (samples will be analyzed in batch at the end of inclusions)
  Number of patients with detected genomic alterations (large rearrangements, LOH and CNV of BRCA1/2 and genes involved in HRD) concordance between DNA extracted from tumour tissue and cfDNA extracted from plasma

CONTACTS AND LOCATIONS:
Overall Officials: GAVOILLE CELINE, MD, Principal Investigator — Institut de Cancérologie de Lorraine; HARLE ALEXANDRE, PhD pharmaD, Study Chair — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France